CLINICAL TRIAL: NCT01056484
Title: Mindfulness Meditation For Alcohol Relapse Prevention
Brief Title: Mindfulness Meditation for Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2009-0118; 1K23AA017508-01A1 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Alcoholism; Substance Use Disorders; Substance Abuse
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Ethanol; Mindfulness; Meditation; Secondary Prevention; Standard of Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation (Experimental): Mindfulness Based Relapse Prevention for Alcohol Dependence intervention + Standard of Care therapy
  Interventions: Behavioral: Mindfulness Based Relapse Prevention for Alcohol Dependence
- Wait-list control (Other): Standard of Care therapy only
  Interventions: Other: "Wait-list" control

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention for Alcohol Dependence — All subjects receive outpatient standard of care (SOC) therapy for alcohol dependence. Experimental subjects also receive the Mindfulness Meditation Relapse Prevention ('meditation') intervention. The intervention is an extension of existing meditation-based therapies for stress, relapse prevention in addictive disorders, and depression. It has been patterned after Mindfulness Based Relapse Prevention and tailored to the specific needs of alcoholics. Its curriculum includes both meditation and "traditional" cognitive therapy relapse prevention components. The intervention consists of an 8-week, manualized meditation course (2 hours/week group sessions) guided by trained instructors. In addition, experimental subjects are asked to meditate at-home (30 min/day, 6 days/week) during the study.
  Other Names: Mindfulness Meditation; Meditation; Mindfulness; Relapse Prevention
  Arms: Meditation
Other: "Wait-list" control — 'Standard of care' (SOC) outpatient therapy for alcohol dependence is provided to all subjects through their outpatient treatment centers and as recommended by their regular providers. Subjects in the control group receive SOC only. Subjects in the experimental arm will receive the study meditation intervention in addition to SOC.
  Other Names: Standard of Care; Treatment as Usual
  Arms: Wait-list control

SUMMARY:
The purpose of this 52-week clinical trial is to see if the meditation-based intervention, adjunctive to standard of care therapy, can reduce relapse and improve psychological health among adults recovering from alcohol dependence.

DETAILED DESCRIPTION:
The goal of this partially-blinded, two-arm clinical trial was to test whether the Mindfulness Meditation Relapse Prevention (meditation), combined with 'standard of care' (SOC) therapy, is more effective in preventing a return to drinking than SOC alone (wait-list control) among adult recovering alcoholics. The intervention was manualized and based on existing models. It was proposed that meditation may improve outcomes of interest through reduction of the severity of stress-related relapse risk factors such as perceived stress, anxiety, depression, craving and emotion dysregulation, and the level of stress-sensitive biomarkers (cytokine interleukin-6, liver enzymes).

For this study, 123 adult alcohol dependent subjects were recruited from collaborating treatment centers, randomly assigned to one of two equal study arms, and followed for 26-weeks (Period 1, Randomized Controlled Trial, RCT). The RCT evaluated the efficacy of the meditation intervention using self-reported alcohol consumption as primary, and drinking-related harms and subject treatment satisfaction and adherence as secondary outcomes. It also gathered preliminary data on potential mechanisms of meditation action. After the completion of their 26-week RCT (Period 1), controls were eligible to receive the meditation intervention ("cross-over"), and all participants were followed-up for additional 26 weeks (non-randomized Period 2).

This study will provide evidence about the efficacy of meditation for alcohol relapse prevention, will further our understanding of relapse and the potential mechanisms of meditation action, direct future research and guide clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence diagnosis
* Completed at least 2 weeks of IOP or (IOP equivalent=at least 2 days per week) for alcohol dependence
* Sober since beginning of outpatient treatment
* English fluency; ability to fill out surveys
* Permanent home address and telephone
* At least 18 years old
* Score >13 on the Perceived Stress Scale

Exclusion Criteria:

* Pregnant
* Alcohol abstinence >14 weeks before enrollment
* Current, regular meditation
* Pre-existing bipolar, schizophrenia, or delusional disorder
* Regular drug use (other than tobacco) in last 2 weeks
* Inability to reliably participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Zgierska, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Background] Zgierska A, Rabago D, Chawla N, Kushner K, Koehler R, Marlatt A. Mindfulness meditation for substance use disorders: a systematic review. Subst Abus. 2009 Oct-Dec;30(4):266-94. doi: 10.1080/08897070903250019. PMID 19904664
- [Background] Zgierska A, Rabago D, Zuelsdorff M, Coe C, Miller M, Fleming M. Mindfulness meditation for alcohol relapse prevention: a feasibility pilot study. J Addict Med. 2008 Sep;2(3):165-73. doi: 10.1097/ADM.0b013e31816f8546. PMID 21768988
- [Background] Marcus MT, Zgierska A. Mindfulness-based therapies for substance use disorders: part 1. Subst Abus. 2009 Oct-Dec;30(4):263-5. doi: 10.1080/08897070903250027. No abstract available. PMID 19904663
- See also: brief description of the findings from the pilot study — http://www.fammed.wisc.edu/research/external-funded/alcohol-prevention

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the initial 26 weeks [Period 1], this was a randomized controlled trial. After the 26 week assessment, control participants were eligible to receive the meditation intervention, however, some elected not to receive the intervention [non-randomized trial]; all study participants were followed up for additional 26 weeks [Period 2].
Groups:
- Meditation: Mindfulness Based Relapse Prevention intervention + Standard of Care therapy
  Mindfulness Based Relapse Prevention for Alcohol Dependence: All study subjects receive outpatient standard of care (SOC) therapy for alcohol dependence. In addition, experimental subjects receive the Mindfulness Meditation Relapse Prevention ('meditation') intervention. This intervention is an extension of existing meditation-based therapies for stress, relapse prevention in addictive disorders, and depression. It has been directly patterned after Mindfulness Based Relapse Prevention and tailored to the specific needs of alcoholics. Its curriculum includes both meditation and "traditional" cognitive therapy relapse prevention components. The intervention consists of an 8-week, manualized meditation course (2 hours/week group sessions) guided by trained instructors. In addition, experimental subjects are asked to meditate at-home (30 min/day, 6 days/week) during the whole study.
Period: Randomized Controlled Trial
Arm/Group | Meditation | Wait-list Control
Started | 64 | 59
Completed | 57 | 58
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Physician Decision | 1 | 0
Period: Follow up - Non-randomized
Arm/Group | Meditation | Wait-list Control
Started | 57 (Out of the enrolled experimental subjects (N=64), 57 completed Period 1 and entered into Period 2.) | 58 (Out of the enrolled control subjects (N=59), 58 completed Period 1 and entered into Period 2.)
Completed | 57 | 56
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meditation | Wait-list Control | Total
Number analyzed (Participants) | 64 | 59 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.1) | 41.9 (11.9) | 41.2 (11.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 59 | 122
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 39 | 31 | 70
Region of Enrollment [Number; unit: participants]
  United States | 64 | 59 | 123

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: Alcohol consumption as measured by percent heavy drinking days from baseline to 26 weeks. A heavy drinking day is defined as 4 or more drinks for women or 5 or more drinks for men, during a 24-hour period.
Time Frame: 26 weeks
Population: Only 105 participants provided data for this measure for the 26-week follow up visit. This was due to participants not providing data as a result of either: declining participation for that visit, being unable to reach within the 26-week follow up time frame, or withdrawing from the study before the 26-week follow up visit.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Meditation | Wait-list Control
Number analyzed (Participants) | 52 | 53
percentage of heavy drinking days | 3.8 (8.4) | 3.0 (8.4)

2. Secondary Outcome: Drinker Inventory of Consequences
Description: Severity of drinking related negative consequences as measured by the Drinker Inventory of Consequences (DrInC-2R). This inventory consists of 50 items rated on a scale of 0 to 3, with '0' indicating a given consequence did not happen, '1' indicating it almost happened, '2' indicating it did happen, and '3' indicating it happened more than once. The sum of all ratings (minus the 5 control questions) indicates the 'total score', with higher scores corresponding to more drinking related consequences. The 'total score' can range from 0 (did not happen) to 135 (happened all the time).
Time Frame: 26 weeks
Population: Only 98 participants provided data for this measure for the 26-week follow up visit. This was due to participants not providing data as a result of either: declining participation for that visit, being unable to reach within the 26-week follow up time frame, or withdrawing from the study before the 26-week follow up visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Meditation | Wait-list Control
Number analyzed (Participants) | 47 | 51
Scores on a scale | 11.3 (16.9) | 16.5 (17.6)

3. Secondary Outcome: Subject Treatment Satisfaction
Description: Treatment satisfaction rating on a Likert scale of 1 to 7 (1 indicating 'extremely dissatisfied', 4 'neutral', and 7 'extremely satisfied').
Time Frame: 8 weeks
Population: 48 participants provided data for this outcome measure at an 8-week follow up visit, and their responses were analyzed.
Measure: Mean (Standard Deviation); unit: points
Groups:
- Meditation: Mindfulness Based Relapse Prevention for Alcohol Dependence intervention
Arm/Group | Meditation
Number analyzed (Participants) | 48
points | 5.5 (1.4)

4. Secondary Outcome: Subject Treatment Adherence
Description: Mindfulness Based Relapse Prevention for Alcohol Dependence intervention session attendance; adherence defined as attending 4 or more out of 8 total sessions.
Time Frame: 8 weeks
Population: Of 64 enrolled participants, one withdrew prior to the first intervention session. This participant's data was included in the baseline data analyses; this participant's meditation intervention attendance was counted as "0".
Measure: Number; unit: Percentage of meditation participants
Arm/Group | Meditation
Number analyzed (Participants) | 64
Percentage of meditation participants | 71.9

5. Primary Outcome: Percent Days Abstinent From Alcohol
Description: Measures percent days abstinent from alcohol
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of days abstinent from alcohol
Arm/Group | Meditation | Wait-list Control
Number analyzed (Participants) | 52 | 53
percent of days abstinent from alcohol | 88.5 (22.5) | 94.1 (11.6)

6. Primary Outcome: Time to Relapse (Resumption of Drinking)
Description: Alcohol consumption as measured by time to relapse (resumption of drinking) from baseline to 26 weeks.
Time Frame: 26 weeks
Population: Only 105 participants provided data for this measure at 26-week follow up; due to participants either: declining participation for the visit, being unable to reach within the 26-week follow up time, or withdrawing from the study before 26-week follow up. Of the 105, 3 meditation/0 controls met criteria for having relapsed during this time frame.
Measure: Mean (Standard Deviation); unit: number of days to relapse
Arm/Group | Meditation | Wait-list Control
Number analyzed (Participants) | 3 | 0
number of days to relapse | 29.0 (13.0) |

ADVERSE EVENTS:
Arm/Group | Meditation | Wait-list Control
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/59
Other Adverse Events (participants affected / at risk) | 0/64 | 0/59

LIMITATIONS AND CAVEATS:
Lack of blinding of study staff to group status (except the statistician who was blinded during initial primary analyses); conducting most study related activities by the same core group of research staff may have introduced bias and placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes